CLINICAL TRIAL: NCT00135070
Title: A Randomised Study Comparing Continuous Intravenous Insulin Infusion With Subcutaneous Insulin Analogues in Hospitalised Patients With Type II Diabetes and Hyperglycaemia
Brief Title: Hospital In-Patient Insulin Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No documentation with MHRA to support clinical trial of a medicinal product.
Sponsor: The Royal Bournemouth Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H.P.I.1
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Detemir

SUMMARY:
Hyperglycaemia has been shown to increase morbidity and mortality in patients with critical illness, myocardial infarction and stroke. This study aims to look at patients with hyperglycaemia and reduce their blood sugar levels using differing combinations of subcutaneous and intravenous insulin.

DETAILED DESCRIPTION:
This is a randomised trial involving patients with type II diabetes who are brought into the hospital with a problem other than a diabetic emergency. Patients will be included, who have a blood sugar > than 17mmols. They will be randomised to one of two groups and either given intravenous or subcutaneous insulin. Outcome measures are length of stay, glucose control and comparison of the two regimens. Cost implications will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes
* Blood glucose > 17mmols

Exclusion Criteria:

* Type I diabetes
* Hyperosmolar non-ketotic coma (HONK)
* Diabetic ketoacidosis (DKA)
* Myocardial infarction (MI)
* Vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Glucose control

SECONDARY OUTCOMES:
Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, Doctor, Principal Investigator — The Royal Bournemouth Hospital
Locations (1):
- The Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom